CLINICAL TRIAL: NCT02438397
Title: Explore the Efficacy of Acarbose and Metformin on Blood Glucose Fluctuation When Combined With Premix Insulin in Chinese Type 2 Diabetes by CGMS
Brief Title: the Efficacy of Acarbose and Metformin on Blood Glucose Fluctuation When Combined With Premix Insulin
Acronym: CGMS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Weiping Jia, Professor,chief of endocrinology department, Shanghai 6th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BHC-17782
Record Dates: First submitted 2015-05-05; First posted 2015-05-08 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin; Metformin; Acarbose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- metformin+premix insulin (Active Comparator): metformin:500mg tid
  Interventions: Drug: premix insulin; Drug: metformin
- acarbose+premix insulin (Experimental): acarbose:100mg tid
  Interventions: Drug: premix insulin; Drug: Acarbose

INTERVENTIONS:
Drug: premix insulin — Premix-insulin(human insulin or analog) treatment will continue
  Other Names: human insulin or analog
Drug: metformin — 500 mg tid by Merck
  Other Names: glucophage
  Arms: metformin+premix insulin
Drug: Acarbose — 100mg tid by Bayer
  Other Names: Glucobay
  Arms: acarbose+premix insulin

SUMMARY:
the study objective: to explore the efficacy of acarbose and metformin on glucose fluctuations as add on therapy in type 2 diabetes patients inadequately controlled with premix insulin.

DETAILED DESCRIPTION:
Study Design:Prospective, parallel group, active-control, randomized, open-label.

Study Organization:Single-center in China. Endocrinology and metabolism department of 6th affiliated hospital of Shanghai Jiaotong university Study Population: Type 2 diabetes inadequately controlled by premix-insulin therapy,40 patients per arm(acarbose add on/ metformin add on) both acarbose and metformin are widely used with premix-insulin in clinical practice, for the better glucose control and lower hypoglycemia incident.

Acarbose delay the absorption of digested carbohydrates from the small intestine and thus lower both postprandial glucose and insulin levels which sequently improve glucose fluctuation Metformin improve the insulin resistance reduce the gluconeogenesis, glucose output and thus lower the fasting glucose

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed T2DM patients (WHO, 1999).
* Premix Insulin therapy for more than 3 months, the daily dosage of insulin >20IU and <1IU/kg
* 30 ≤Age ≤ 70 years old, male or female
* 7.0 ≤ HbA1c ≤10.0%
* 18.5≤ BMI ≤ 35 kg/m2
* Written Informed consent

Exclusion Criteria:

* Subject with type 1 diabetes or gestational diabetes mellitus and other specific types DM
* Those who can not tolerate AGI or who is suffering GI disease
* Metformin contradiction
* Concomitant 2 oral anti-diabetes medicine, or 1 OAD with maximum dose
* Subject with repeated severe hypoglycemia and/or unawareness of hypoglycemia
* Known or suspected allergy to trial product(s) or related products
* Females of child bearing potential who are pregnant, breast-feeding or have the intention of becoming pregnant or not using adequate contraceptive methods throughout the trial
* Impaired liver function,
* Any other clinically significant condition or major systemic diseases, including serious coronary heart disease, cardiovascular disease, cancer, TB, acute infection
* Uncontrolled hypertension
* Concomitant treatment which influences blood glucose
* Impaired renal function

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
MAGE: mean amplitude of glycemic excursion/MODD: mean of daily differences | 12 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Weiping Jia, doctor, Principal Investigator — the 6th affiliated hospital of Shanghai Jiaotong university
Locations (1):
- the 6th affliliated hospital of Shanghai Jiaotong university, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Gao F, Li C, Wang Y, Lu J, Lu W, Zhou J, Yin J, Ma X. Growth differentiation factor 15 is not associated with glycemic control in patients with type 2 diabetes mellitus treated with metformin: a post-hoc analysis of AIM study. BMC Endocr Disord. 2022 Oct 22;22(1):256. doi: 10.1186/s12902-022-01176-3. PMID 36273168